CLINICAL TRIAL: NCT03698006
Title: Optimal Pain Control After Prothetic Knee Surgery Either by Selective Tibial Nerve Block Versus Local Infiltration Analgesia
Brief Title: Selective Tibial Nerve Block vs Local Infiltration Analgesia After Prothetic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2018-01080
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain; Knee Osteoarthritis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibial nerve block (Experimental): Adductor canal and tibial nerve blocks performed by the anesthetist under ultrasound guidance before spinal block.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- Local infiltration analgesia (Active Comparator): Adductor canal block by the anesthetist under ultrasound guidance before spinal block. Infiltration of the knee by the surgeon with local anesthetic at the end of the surgery.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Tibial nerve block with 10ml of Ropivacaine 0.5%
  Arms: Tibial nerve block
Drug: Ropivacaine 0.2% Injectable Solution — Infiltration with 25ml of Ropivacaine 0.2% in the posterior knee capsule
  Arms: Local infiltration analgesia

SUMMARY:
Patient suffer from moderate posterior knee pain after TKA despite injection of local anesthetic around the femoral or saphenous nerves. Indeed, the posterior part of the knee is innervated by the sciatic nerve. This nerve is not routinely blocked as clinicians fear to produce a motor block of the leg that might impair the postoperative assessment. An analgesic alternative is the infiltration of the knee with local anesthetics performed by the surgeon. Recently a trial(1) demonstrated that a selective tibial nerve block provides an effective analgesia without a motor blockage when compared with a sciatic nerve block. The objective of this randomized controlled double-blinded trial is to assess whether a tibial nerve block is more effective for the postoperative pain than local infiltration analgesia when there are combined with an adductor canal block, without decreasing the functional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for a total knee arthroplasty under spinal block.
* Patient with a weight above 40kg.

Exclusion Criteria:

* Patient with ASA IV status.
* Contraindication to spinal block, or peripheral nerve blocks.
* Neurological deficit of the lower limb.
* Patient with renal dysfunction.
* Patient with chronic pain, opioid consumption or alcohol consumption.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption (mg) | 24 hours postoperatively

SECONDARY OUTCOMES:
Total morphine consumption (mg) | 2 hours, 48 hours and 72 hours postoperatively
Analgesic duration (minutes) | Postoperative day 0
  Time from the block to the first analgesic request
Pain scores (numeric rating scale, 0-10) at rest and on movement | 2 hours, 24 hours, 48 hours and 72 hours postoperatively
  0= no pain, 10=the worst pain imaginable
Rate of postoperative nausea and vomiting | 2 hours, 24 hours, 48 hours and 72 hours postoperatively
  Yes/No
Rate of prurit | 2 hours, 24 hours, 48 hours and 72 hours postoperatively
  Yes/No
Active flexion | 24hours, 48hours and 72hours postoperatively
  Flexion of the knee by the patient measured in degrees
Passive flexion | 24hours, 48hours and 72hours postoperatively
  Flexion of the knee by physiotherapist measured in degrees
Quadriceps muscle strength (numeric scale, 1-5) | 24hours, 48hours and 72hours postoperatively
  1=no contraction, 5=normal strength
Distance walked (meters) | 24hours, 48hours and 72hours postoperatively
Complication of tibial nerve block | up to 1 week
  Intravascular injection/hematoma/infection/Common peroneal nerve block
Length of stay in hospital | up to 14 days
  Days

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Albrecht, Lausanne, English, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinha SK, Abrams JH, Arumugam S, D'Alessio J, Freitas DG, Barnett JT, Weller RS. Femoral nerve block with selective tibial nerve block provides effective analgesia without foot drop after total knee arthroplasty: a prospective, randomized, observer-blinded study. Anesth Analg. 2012 Jul;115(1):202-6. doi: 10.1213/ANE.0b013e3182536193. Epub 2012 Apr 27. PMID 22543069